CLINICAL TRIAL: NCT05122390
Title: Can a Mobile Application, Contraction Coper, Better Prepare Women in Early Labour and Reduce Emotional Distress for Nulliparous Women? A Randomised Control Trial (the Digi-EL Trial) in a Swedish Sample
Brief Title: DIGItal Early Labour. A Digital Application for Coping in Early Phase of Labour.
Acronym: DIGI-EL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Värmland County Council, Sweden (Other Government)
Collaborators: Karlstad University (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CcVarmland
Record Dates: First submitted 2021-09-23; First posted 2021-11-16 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy Related
Keywords: emotional distress; digital application

STUDY DESIGN:
Intervention Model Description: The experimental group is divided into two groups, one group that gets access to the application Contraction Coper only and one group gets Contraction Coper Plus, both the application and additional support of the midwife through blended care. The third group is standard care only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contraction Coper (Experimental): The digital application Contraction Coper is provided from pregnancy week 25. The application contains two different modules. One is an informational module about the method (about 60 minutes), the other is a contraction module to be used in early labour (in total 6 hours).
  Interventions: Other: Contraction Coper
- Contraction Coper Plus (Active Comparator): The digital application Contraction Coper with additionally support from a midwife in two different occasions during pregnancy.
  Interventions: Other: Contraction Coper; Other: Contraction Coper Plus
- Control (No Intervention): Conventional antenatal care.

INTERVENTIONS:
Other: Contraction Coper — Digital application built on the Birth without fear method, based on four different tools to be used during labour. Breathing, relaxation, voice and mind.
  Arms: Contraction Coper; Contraction Coper Plus
Other: Contraction Coper Plus — Digital application built on the Birth without fear method, based on four different tools to be used during labour. Breathing, relaxation, voice and mind. Clinical guidance from a midwife during two different occasions is added to the group.
  Arms: Contraction Coper Plus

SUMMARY:
All first-time mothers in Sweden are offered parental support, but local conditions mean that not everyone gets the opportunity to take part in this. Studies show that there is a lack of evidence-based guidelines for the design of parental support in maternal health care. Early labour or latent phase of labour is the part of childbirth were women often feel insecure, in stress and left out from care. First-time mothers who have no experience of one labour before are particularly vulnerable. Many women today use digital applications during pregnancy and in connection with childbirth. There are several digital applications that will help the woman by guiding her and her partner in different decisions about labour, but it is necessary to offer evidence-based, credible electronic and digital solutions for expectant parents. A meta-synthesis from 2018 showed that women use the internet often and the information they receive there has a great influence on their different choices in connection with childbirth. Volume, accessibility, and convenience about digital solutions play a crucial role for women and partners. The digital application Contraction Coper is designed and tested by the company Birth By Heart © in order to facilitate in early labour for the pregnant woman and her partner. The overall purpose of the project is to evaluate whether the application Contraction Coper can contribute to reduced anxiety and stress during pregnancy and childbirth and whether an additional support from a midwife can increase the application use and satisfaction of women when using the application.

A randomized controlled trial is planned where first-time mothers after pregnancy week 25 are invited to participation via social platforms. Participating first-time mothers are randomly assigned to one of three groups; experiment group one, which gets access to the application Contraction Coper, experiment group two Contraction Coper Plus which gets access to both the application and support of midwives, so-called "blended" care, or three, the control group offered customary maternity care only.

Data collection is conducted using questionnaires, mobile application and activity bracelet.

DETAILED DESCRIPTION:
The primary outcome is emotional stress in early labour measured with the dimension "Emotional Distress" in the questionnaire Early Labour Experience Questionnaire (ELEQ) Secondary outcomes are Fear of Birth Scale(FOBS), Childbirth Experience Questionnaire (CEQ), used pain relief methods during labour and birth, mode of birth, amount of time used in the application as well as heart rate, sleep and activity for the experimental groups that had activity bracelets in addition.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers
* From pregnancy week 25.
* Swedish or English spoken.
* Having a Smartphone, Android or Apple application.

Exclusion Criteria:

°Multiparas.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant persons
Enrollment: 480 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Emotional distress | "Group differences at 1 month after birth"
  The subscale Emotional distress from Early Labour Experience Questionnaire (ELEQ) will be used for measure. Emotional distress scale is assessed on a five point Likert scale 1-5. Minimum score 6 and maximum score is 30. A higher score represents more distress during early labour.

SECONDARY OUTCOMES:
Fear of birth | "Assesed during pregnancy week 25 up till week 36 at consent to the study"
  Fear of forthcoming birth will be measured with Birth scale (FOBS) by a question 'How do you feel right now about the approaching birth?' by placing a mark on two different 10-cm lines, by using the anchors; (a)'calm' and 'worried' and (b) 'no fear' and 'strong fear' creating an average of minimum score is 0 and maximum score 100 with high scores indicating higher levels of childbirth fear. Cut off point is considered at 60.
Fear of birth in potential future birth | " Group differencies at 1 month after birth"
  Fear of Birth scale (FOBS) will be used and asked by a question 'How do you feel right now about a potential future birth?' by placing a mark on two different 10-cm lines, by using the anchors; (a)'calm' and 'worried' and (b) 'no fear' and 'strong fear' creating an average of minimum score is 0 and maximum score 100 with high scores indicating higher levels of childbirth fear. Cut off point is considered at 60. Pairwise analyse with score before birth.
Sense of coherence | "Assessed during pregnancy week 25 up till week 36 at consent to the study"
  Sense of Coherence will be measured with SOC-13 (short version). Each question is answered between 1-7. The summed score ranges between 13 and 91. Score is categorized into low(<60), moderate (61-75) and high (>76) SOC.
Childbirth experience | "Group differencies at 1 month after birth"
  Childbirth Experience Questionnaire(CEQ) will be used. The questionnaire contains four different dimensions. The items (n=22) are measured on a four point Likert scale. Minimum is 22 and maximum 88. A higher value represents a more positive chidbirth experience.
Support from birth companion | "Group differencies at1 month after birth"
  The Birth Companion Support Questionnaire (BCSQ) will be used for measuring the support the woman experiences from her partner during labour and birth and contains two different dimensions. 12 items are answered on a 4 point Likert scale. Minimum is 12 and maximum is 48. A higher score represents a more positive attitude about recieved support.
Childbirth Self-Efficacy Inventory before childbirth | "Assessed during pregnancy week 25 up till week 36 at consent to the study"
  The Swedish version of Child Birth Self-efficacy Inventory, (CBSEI) will be used. The questionnaire measuring self-efficacy on both outcome expectancies, i.e. 'what behavior do you think would be useful during labour' as well as self-efficacy expectancies, i.e.' how do you think you will be able to conduct yourselves during labour'. The 15 questions will be asked on ten point Likert scale. ranging from 1 to 10; higher scores indicate a higher degree of childbirth self-efficacy. Minimumscore is 15 and maximum scores are 150 on both scales.
Childbirth Self-Efficacy Inventory after childbirth | "Group differencies at1 month after birth"
  The Swedish version of Child Birth Self-efficacy Inventory (CBSEI) with the assessment of self-efficacy after childbirth. 'How did you conduct yourselves during labour'. The 15 questions will be asked on ten point Likert scale. ranging from 1 to 10; higher scores indicate a higher degree of childbirth self-efficacy during childbirth. Minimumscore is 15 and maximum scores are 150. Pairwise analysis with score before birth for analysis.
Activity bracelet FitBit | "At the timepoint were contractions starts during early labour and until the baby is born"
  Heartrate is measured using activity bracelet. A higher heartrate indicates more pain and distress
Activity bracelet FitBit | "At the timepoint were contractions startsduring early labour and until the baby is born"
  Sleep pattern is measured using activity bracelet. A shorter and interrupted sleep indicates more pain and distress

OTHER OUTCOMES:
Labour outcome from medical record | "At birth"
  Mode of birth; vaginal, vaccuum extraction, cesarean section
Medical interventions during labour from medical record | "During labour and birth"
  Amniotomy, oxytocin augmentation yes/no
Length of labour phases from medical record | "During labour and birth"
  Length of latent phase, length of active phase, length of pushing phase, measured in minutes and hours
Pain relif methods used from medical record | "During labour and birth"
  Nitrus oxide, Epidural, Spinal, non-medical pain relief yes/no
Apgar Score from medical record | "At birth and during first week after birth"
  Apgar Score ranging from 1-10, at 1 and 5 and 10 minutes after childbirth. Minimum 0-0-0 and maximum 10-10-10.
Neonatal outcome from medical record | "At birth and during first week after birth"
  Neonatal care at neonatal intensive unit within one week after childbirth, yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ängeby, PhD, Principal Investigator — Region Värmland
Locations (2):
- Sweden (2):
  - Women's department, Karlstad
  - County of Värmland, Karlstad

IPD SHARING:
Plan to Share IPD: No